CLINICAL TRIAL: NCT03819933
Title: Optimizing Family Counseling for Anticipated Extremely Preterm Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); South Shore Hospital (Other)
Responsible Party: Principal Investigator, Christy Cummings, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB-P00030146
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Preterm Pregnancy; Premature Birth
Keywords: Counseling; Extreme Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This pre/post, mixed method behavioral intervention study will enroll ~130 families (pregnant women and their partners) at extreme prematurity and their counseling providers from Maternal Fetal Medicine (MFM) and Neonatology (total possible participants ~460) to determine whether developed educational interventions for providers (workshop, online module or both) improve counseling practices and outcomes using comparative statistical analyses.
Masking Description: There will be no masking in this behavioral intervention trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women and their partners (Other): For the qualitative arm of this mixed method study, using an exploratory sequential design, investigators will enroll ~ 30 adult pregnant women admitted estimated 22 0/7-25 6/7 weeks' estimated gestation and their partners to participate in a post-counseling semi-structured interview to explore preferred language and approaches, and better inform questionnaire development. Sample size will be up to 30 families, or until thematic saturation is achieved (total up to 60 if all partners agree to participate).
  For the quantitative arm of this study, investigators will enroll ~100 adult pregnant women admitted between estimated 22 0/7-25 6/7 weeks' estimated gestation and their partners (up to total ~200 if all partners present and agree to participate).
  Interventions: Behavioral: Educational intervention
- Counseling MFM and Neonatology providers (Other): Investigators will enroll ~100 counseling Maternal-Fetal Medicine (MFM) specialists and 100 counseling Neonatologists (total ~200 providers), who provided counseling to the enrolled pregnant women between 22 0/7-25 6/7 weeks' estimated gestation for anticipated extremely preterm delivery. This assumes 1 counseling provider from MFM and 1 from Neonatology per pregnant woman, although there could be more if a consult is performed by both an attending physician and a training fellow or practitioner, or less, if a counseling provider declines to participate in the study. There will be anticipated repetition of counseling providers, accounted for in the statistical analysis. Providers will be asked to complete educational interventions to improve counseling at extreme prematurity.
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — Investigators will first determine preferred language and approaches by families, then redefine current training for prenatal counseling at extreme prematurity by developing and implementing two novel, interdisciplinary simulation-based educational programs for MFM and Neonatology (a workshop and an online module), focusing on eliciting values and building partnerships through advanced communication and relational skills, to improve counseling practices and outcomes

SUMMARY:
Antenatal family counseling for anticipated extremely preterm deliveries remains ethically and practically challenging for maternal-fetal medicine specialists and neonatologists alike. The overall goal of this project is to improve antenatal counseling and counseling outcomes for families facing anticipated extremely preterm delivery through innovative, interdisciplinary simulation-based education for maternal fetal medicine specialists and neonatologists, using language preferred by families, and focusing on eliciting values and building partnerships through advanced communication and relational skills.

DETAILED DESCRIPTION:
Extremely preterm birth near the limit of viability, defined broadly as birth between 20 and 26 weeks' gestation, accounts for substantial infant morbidity and mortality as well as both parental and provider distress. Prenatal counseling for families anticipating extremely preterm delivery remains ethically and practically challenging for both Maternal Fetal Medicine (MFM) specialists and neonatologists. Physicians must quickly establish a trusting relationship with families and convey complex medical information. They must sensitively elicit family preferences and values regarding life and death, carefully explain management options and potential outcomes such as long-term disability, and arrive at a mutually agreeable plan for delivery and resuscitation. However, prenatal counseling may be disjointed or even contradictory. It has been shown that suboptimal counseling is partially explained by differences in training, practice and perspectives between the specialties, as well as in framing and unconscious biases, time constraints and poor communication. Physicians also often emphasize cognitive information versus parental values when counseling. Preferred language and counseling approaches are largely unknown. This can lead to poor family understanding, inadequate shared decision making, decreased satisfaction and increased anxiety.

There is a need to determine best approaches using language and terminology preferred by families, not physicians. There is also a need to develop new methods to educate MFM and Neonatology providers to improve antenatal counseling. Simulation and enactments are effective in teaching patient-physician communication, ethical dilemmas in medicine, and prenatal counseling. This mixed-methods behavioral intervention study will first determine preferred language and approaches by families, then redefine current training for prenatal counseling at extreme prematurity by developing and implementing two novel, interdisciplinary simulation-based educational programs for MFM and Neonatology, focusing on eliciting values and building partnerships through advanced communication and relational skills, to improve counseling practices and outcomes.

The overall hypothesis is that family-focused counseling at extreme prematurity by providers trained in using language and approaches preferred by families will more effectively address parents' values and preferences central to decision making and improve counseling practices and outcomes. In this mixed-methods study, the investigators will enroll ~130 families and their counseling providers from MFM and Neonatology and compare family-focused counseling outcomes after educational interventions to baseline. Investigators will collaborate with Family Faculty advisors from study design through publication to incorporate the parental perspective.

Aim 1a: To determine, via semi-structured interviews of up to 30 families, preferred language, terminology and approach, including maternal/paternal differences, during family counseling for impending extremely preterm delivery, following standard counseling. Aim 1b: To establish baseline understanding, perceptions, decision making, and anxiety of 50 families and their counseling providers measured via survey, including the Controlled Preferences Scale-Pediatrics, Decisional Conflict Scale, and State Trait Anxiety Inventory (STAI). Secondary hypothesis: maternal/paternal preferences for language, involvement and decision making differ.

Aim 2a: To develop a novel, joint-specialty simulation-based workshop for MFMs and neonatologists through Boston Children Hospital's (BCH) established Simulation Pediatric Program and Institute for Professionalism and Ethical Practice (IPEP). Aim 2b: To create an innovative, multi-media online training module for MFMs and neonatologists through BCH Simulation Pediatric/IPEP and Open PediatricsTM, a free and globally accessible web-based teaching platform to enable widespread dissemination. Both products will use preferred language and approaches from a national survey by investigators (in progress) and Aim 1, while emphasizing interdisciplinary communication, ethical and relational skills, addressing biases, and focusing on family values and preferences central to decision making.

Aim 3: To evaluate whether developed educational interventions improve counseling practices and outcomes on repeat surveys of 50 families and trained counseling providers using comparative statistical analyses. Primary hypothesis: counseling by trained providers will improve parental 1) understanding, 2) perceptions, 3) decision making, and 4) anxiety, by improving communication and more effectively addressing parents' values and preferences central to decision making. Secondary hypotheses: 1) the online module will be as effective as the workshop; 2) trained providers will report increased comfort and decreased anxiety when counseling.

Given the weight of decisions resulting from family counseling for impending extremely preterm delivery, joint-specialty interventions using preferred language and approach to optimize counseling are urgently needed. These innovative educational interventions present a feasible and effective approach that can be widely disseminated to improve interdisciplinary family-focused counseling for anticipated extremely preterm deliveries and counseling outcomes, representing a direct and immediate clinical impact.

ELIGIBILITY:
1. Pregnant women and their partners

   Inclusion Criteria:
   * English-proficient adult pregnant woman admitted between 22 0/7-25 6/7 weeks' estimated gestation for anticipated extremely preterm delivery and her adult partner (if available) for whom an antenatal neonatal intensive care unit (NICU) consultation was requested and performed

   Exclusion Criteria:
   * Non-English proficient
   * Fetal congenital malformation(s)
   * <18y old
   * <22 0/7 or > 25 6/7 weeks' estimated gestation
   * Repeat consultation
2. Counseling MFM and Neonatology providers

Inclusion Criteria:

* Practicing MFM or Neonatology provider (attending, fellow, resident, practitioner or RN) from the 3 participating sites: Brigham & Women's Hospital (BWH), Beth Israel Deaconess Medical Center (BIDMC), South Shore Hospital (SSH)

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Parental knowledge | 5 years
  The Parental Questionnaire includes questions asking about parental knowledge and understanding about extremely preterm deliveries and clinical outcomes post-counseling to assess parental knowledge and compare pre/post educational interventions. Question format includes Yes/No (which will be averaged and compared pre/post), 5-point Likert scales (ranging "Not at all" to "Extremely" for various topics) as well as free text boxes for qualitative analyses. Likert scale responses will be collapsed into 2 or 3 levels for analyses.
Parental satisfaction: The Parental Questionnaire | 5 years
  The Parental Questionnaire includes questions asking about parental satisfaction and perceptions post-counseling to compare pre/post educational interventions. Question format includes Yes/No (which will be averaged and compared pre/post), 5-point Likert scales (ranging "Not at all" to "Extremely" for various topics) as well as free text boxes for qualitative analyses. Likert scale responses will be collapsed into 2 or 3 levels for analyses.
Parental decision making | 5 years
  The Parental Questionnaire includes the Controlled Preferences Scale-Pediatrics (CPS-P) and the Ottawa Decisional Conflict Scale (ODCS) to assess parental decision making and compare pre/post educational interventions. The CPS-P is a validated, reliable tool adapted for use in pediatrics to assess parental preferences for participation in decision making and consists of 5 statements describing various roles in decision making, ranging from passive ("I prefer to leave all decisions regarding my child's treatment to my doctor") to active ("I prefer to make the final decision about which treatment my child will receive"), to collaborative. The ODCS is a validated 16-item tool with 5 response categories that measures personal perceptions of decision making. Each of the 16 DCS items is given a score value ranging 0-4, which are summed, divided by 16, and multiplied by 25, yielding a total score ranging from 0-100 (no decisional conflict - extremely high decisional conflict).
Parental anxiety | 5 years
  The Parental Questionnaire includes the State Trait Anxiety Inventory (STAI) to assess parental anxiety and compare pre/post educational interventions. The Spielberger State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait (baseline) and state (present) anxiety, used in clinical research to detect patient and caregiver changes in state of anxiety.58-61 In the third section of the Parental Questionnaire, participants will be asked 20 questions from the STAI, which is appropriate for participants with at least a 6th grade reading level, to measure current levels of anxiety, as opposed to a tendency towards anxiety at baseline. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." All items are rated on a 4-point scale, ranging from "Almost Never" to "Almost Always," with higher scores indicating greater anxiety.
Parental preferred language and terminology | 5 years
  The Parental Questionnaire includes questions asking about preferred parental language and terminology when counseling at extreme prematurity. Question format includes Yes/No (which will be averaged and compared pre/post), 5-point Likert scales (ranging "Not at all" to "Extremely" for various topics) as well as free text boxes for qualitative analyses. Likert scale responses will be collapsed into 2 or 3 levels for analyses.

SECONDARY OUTCOMES:
Maternal versus Paternal/Partner preferences | 3 years
  The Parental Questionnaire includes questions asking about parental preferences for language, involvement and decision making at extreme prematurity, including the CPS-P and ODCS (see above), to detect any maternal versus paternal/partner differences. Question format includes Yes/No (which will be averaged and compared pre/post), 5-point Likert scales (ranging "Not at all" to "Extremely" for various topics) as well as free text boxes for qualitative analyses. Likert scale responses will be collapsed into 2 or 3 levels for analyses.
Effect of Educational Interventions | 2 years
  The Parental and Provider Questionnaires include questions asking about parental and provider knowledge, satisfaction, decision making, anxiety (tools described above) regarding counseling at extreme prematurity to determine whether developed educational interventions for providers (workshop, online module or both) improve counseling practices and outcomes using comparative statistical analyses. Question format includes Yes/No (which will be averaged and compared pre/post), 5-point Likert scales (ranging "Not at all" to "Extremely" for various topics) as well as free text boxes for qualitative analyses. Likert scale responses will be collapsed into 2 or 3 levels for analyses.
Provider anxiety | 5 years
  The Provider Questionnaire includes the State Trait Anxiety Inventory (STAI) to assess provider anxiety when counseling at extreme prematurity and compare pre/post educational interventions. The Spielberger State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait (baseline) and state (present) anxiety, used in clinical research to detect patient and caregiver changes in state of anxiety.58-61 In the third section of the Parental Questionnaire, participants will be asked 20 questions from the STAI, which is appropriate for participants with at least a 6th grade reading level, to measure current levels of anxiety, as opposed to a tendency towards anxiety at baseline. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." All items are rated on a 4-point scale, ranging from "Almost Never" to "Almost Always," with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Christy Cummings, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Boston Children's Hosptial, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts